CLINICAL TRIAL: NCT04493411
Title: Noninvasive Detection and Assessment of Therapy Response in Multiple Myeloma Using Whole-Body MRI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding expired before enrollment goal could be reached.
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Avneesh Chhabra, Professor, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STU-2019-0834
Record Dates: First submitted 2020-07-23; First posted 2020-07-30 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Multiple Myeloma
Keywords: magnetic resonance imaging; positron emission tomography
MeSH Terms: conditions — Multiple Myeloma | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Multiple Myeloma Patients (Experimental): Patients with pathologically confirmed myeloma for cross-sectional study (detection) or scheduled to undergo induction therapy (or have gone 1-2 cycles of induction therapy), followed by either bone marrow transplantation or consolidation therapy for longitudinal study (therapy response assessment).
  Interventions: Procedure: WBMRI; Procedure: Positron Emission Tomography/Computed Tomography (PET/CT)

INTERVENTIONS:
Procedure: WBMRI — WBMRI will be performed either at 1 time point for cross-sectional study or at 4 timepoints for the longitudinal study at the following time points.
  1. Baseline: (before or after 1-2 cycles of induction therapy)
  2. Between Week 12 - 24 (before Bone Marrow Transplant or undergoing consolidation therapy)
  3. Between Week 24 - 36 (before starting maintenance therapy)
  4. Between Week 60 - 72 (post bone marrow transplant or consolidation therapy and after approximately 9 months of maintenance therapy)
Procedure: Positron Emission Tomography/Computed Tomography (PET/CT) — PET/CT will be performed at at 1 time point for cross-sectional study or at 4 timepoints for the longitudinal study at the following time points.
  1. Baseline: (before or after 1-2 cycles of induction therapy)
  2. Between Week 12 - 24 (before Bone Marrow Transplant or undergoing consolidation therapy)
  3. Between Week 24 - 36 (before starting maintenance therapy)
  4. Between Week 60 - 72 (post bone marrow transplant or consolidation therapy and after approximately 9 months of maintenance therapy)

SUMMARY:
This study is designed to prospectively determine the sensitivity, specificity, and diagnostic accuracy of whole-body MRI (WBMRI) with Dual-Echo T2-weighted acquisition for Enhanced Conspicuity of Tumors (DETECT) for the detection of multiple myeloma.

Subjects will undergo WBMRI and fluorodeoxyglucose (FDG) positron emission tomography (PET) for research purposes either at one time point for cross-sectional study or at four time points for longitudinal study: baseline, prior to bone marrow transplant (BMT), prior to maintenance therapy, and post BMT. The results of these imaging procedures will be compared to standard of care whole body x-ray and bone marrow biopsy results.

DETAILED DESCRIPTION:
Whole body magnetic resonance imaging (WBMRI) will be evaluated for detection and assessment of therapy response in multiple myeloma (MM) using a novel acquisition scheme. WBMRI with diffusion weighted imaging (DWI) has demonstrated promising preliminary results for detection and response monitoring in MM. While DWI generates high lesion-to-background contrast and excellent lesion conspicuity, it suffers from compromised image quality due to geometric distortion, particularly at 3 Tesla magnetic resonance imaging (MRI), a platform which is increasingly used in clinical practice. This disadvantage, along with high costs and patient dissatisfaction associated with long scan times, have limited wide spread adoption of WBMRI with DWI in the clinical practice.

To overcome these challenges, the investigators have developed an alternative WBMRI technique: Dual-Echo T2-weighted acquisition for Enhanced Conspicuity of Tumors (DETECT) for improved tumor visualization by simultaneously suppressing the confounding signals of fat and fluid throughout the body.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pathologically confirmed myeloma.
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0, 1, or 2.
* For cross-sectional study, no additional required treatment schedule. For longitudinal study: Patients scheduled to undergo bone marrow biopsy (BMB) and induction therapy (or have gone through 1-2 cycles of induction therapy), followed by either bone marrow transplantation (BMT) or consolidation therapy.
* Women of child-bearing potential must agree to undergo a urine pregnancy screening to prevent imaging of pregnant patients. A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria: 1) Has not undergone a hysterectomy or bilateral oophorectomy; or 2) Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).
* Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

* Subjects may not be receiving any other investigational agents for the treatment of the cancer under study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that, in the opinion of the investigator, would limit compliance with study requirements.
* Subjects must not be pregnant or nursing; since pregnancy is a contraindication to administration of gadolinium-based contrast agents. Furthermore, there is a potential for congenital abnormalities and the potential to harm nursing infants, associated with FDG-PET.
* Any contraindication to MRI per Radiology Department's routine protocol, e.g. MRI-incompatible objects, including but not limited to medical devices and other foreign bodies.
* Known severe allergic reaction to Gadolinium-based contrast agents.
* Patients with uncontrollable claustrophobia, severe lower back pain, and uncontrollable tremors, to the point that it would render them unable to tolerate an MRI study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2024-04-12 (Actual); Study Completion 2024-04-12 (Actual)

PRIMARY OUTCOMES:
Detection of lesions | Up to 4 years
  Effectiveness of WBMRI DETECT for the detection of lesions in MM patients will be compared to WBMRI Diffusion Weighted Imaging (DWI). A combination of clinical MRI, whole body x-ray, FDG PET, and bone marrow biopsy will be used as the reference standard.
  The number of lesions identified on WBMRI-DETECT will be compared to the number of lesions identified on WBMRI-DWI. The sensitivity and specificity of WBMRI-DETECT and WBMRI-DWI will be calculated using the reference standard.
Assessment of therapy response | Up to 4 years
  Effectiveness of WBMRI for assessing therapy response will be compared to the current standard of care using FDG PET and bone marrow biopsy as the validation standard.
  The percentage increase in fat fraction measured using WBMRI-DETECT and the percentage increase in apparent diffusion coefficient (ADC) measured using WBMRI-DWI will be used to assess the effectiveness of WBMRI in measuring therapy response. The percentage change in SUVmax measured on PET/CT will be used as the reference standard.
Progression Free Survival (PFS) | Up to 4 years
  Will determine if WBMRI prognosis is at baseline, after 4-6 weeks of induction therapy, and before maintenance therapy is associated with PFS.
Overall Survival (OS) | Up to 4 years
  Will determine if WBMRI prognosis is at baseline, after 4-6 weeks of induction therapy, and before maintenance therapy is associated with OS.

CONTACTS AND LOCATIONS:
Overall Officials: Avneesh Chhabra, MD, PhD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No